CLINICAL TRIAL: NCT00905645
Title: Sientra Sponsored Silimed Gel-Filled Mammary Implant Clinical Study Protocol: Core Clinical Investigation
Brief Title: Sientra Sponsored Silimed Gel-Filled Breast Implant Core Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tiger Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G010193
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-09

CONDITIONS: Breast Augmentation; Breast Reconstruction; Breast Revision
Keywords: Breast Augmentation; Breast Reconstruction; Breast Revision; Silicone breast implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Primary Augmentation (Experimental): Silimed Gel-Filled Mammary Implant
  Interventions: Device: Silimed Gel-Filled Mammary Implant
- Revision-Augmentation (Experimental): Silimed Gel-Filled Mammary Implant
  Interventions: Device: Silimed Gel-Filled Mammary Implant
- Primary Reconstruction (Experimental): Silimed Gel-Filled Mammary Implant
  Interventions: Device: Silimed Gel-Filled Mammary Implant
- Revision-Reconstruction (Experimental): Silimed Gel-Filled Mammary Implant
  Interventions: Device: Silimed Gel-Filled Mammary Implant

INTERVENTIONS:
Device: Silimed Gel-Filled Mammary Implant

SUMMARY:
Safety and effectiveness of the Silimed Gel-Filled Mammary Implant as indicated for primary augmentation, primary reconstruction, and/or revision of the female breast.

ELIGIBILITY:
Inclusion Criteria

Subjects are admitted into the study only if all of the following eligibility is true:

* Female
* Age limitation specific to the indication:

  * Primary Augmentation: Must be 18 years or older
  * Primary Reconstruction: No age limit
  * Revision: If original surgery was primary reconstruction, then no age limit. If original surgery was primary augmentation, then must be 18 years or older.
* Adequate tissue available to cover implant(s)
* Willingness to follow study requirements (informed consent form, follow-up visits)
* Candidate for primary augmentation, primary reconstruction, or revision

Exclusion Criteria

Subjects are not eligible if any of the following criteria exist:

* Advanced fibrocystic disease, considered to be pre-malignant without mastectomy
* Inadequate or unsuitable tissue
* Active infection in the body at the time of surgery
* Pregnant or lactating
* Medical condition that might result in unduly high surgical risk and/or significant postoperative complications, in the judgment of the Investigator
* Use of drugs, including any drug that would interfere with blood clotting, that might result in high risk and/or significant postoperative complications
* Demonstrated psychological characteristics that are unrealistic or unreasonable given the risks involved with the surgical procedure
* Determination by physical examination that the subject does have any connective tissue/autoimmune disorder
* Existing carcinoma of the breast without accompanying mastectomy
* MRI scan is prohibited because of implanted metal device, claustrophobia, or other condition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1788 (Actual)
Dates: Start 2002-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Dajles, PhD, Study Director — Tiger Biosciences, LLC.
Locations (1):
- Sientra, Inc., Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevens WG, Harrington J, Alizadeh K, Berger L, Broadway D, Hester TR, Kress D, d'Incelli R, Kuhne J, Beckstrand M. Five-year follow-up data from the U.S. clinical trial for Sientra's U.S. Food and Drug Administration-approved Silimed(R) brand round and shaped implants with high-strength silicone gel. Plast Reconstr Surg. 2012 Nov;130(5):973-981. doi: 10.1097/PRS.0b013e31826b7d2f. PMID 23096598
- [Background] Stevens WG, Harrington J, Alizadeh K, Broadway D, Zeidler K, Godinez TB. Eight-year follow-up data from the U.S. clinical trial for Sientra's FDA-approved round and shaped implants with high-strength cohesive silicone gel. Aesthet Surg J. 2015 May;35 Suppl 1:S3-10. doi: 10.1093/asj/sjv020. PMID 25948657
- [Background] Stevens WG, Calobrace MB, Harrington J, Alizadeh K, Zeidler KR, d'Incelli RC. Nine-Year Core Study Data for Sientra's FDA-Approved Round and Shaped Implants with High-Strength Cohesive Silicone Gel. Aesthet Surg J. 2016 Apr;36(4):404-16. doi: 10.1093/asj/sjw015. PMID 26961987
- [Background] Stevens WG, Calobrace MB, Alizadeh K, Zeidler KR, Harrington JL, d'Incelli RC. Ten-year Core Study Data for Sientra's Food and Drug Administration-Approved Round and Shaped Breast Implants with Cohesive Silicone Gel. Plast Reconstr Surg. 2018 Apr;141(4S Sientra Shaped and Round Cohesive Gel Implants):7S-19S. doi: 10.1097/PRS.0000000000004350. PMID 29595714

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Augmentation | Revision-Augmentation | Primary Reconstruction | Revision-Reconstruction
Started | 1116 | 363 | 225 | 84
Completed | 688 | 192 | 118 | 32
Not Completed | 428 | 171 | 107 | 52
Not completed — Death (not device related) | 10 | 4 | 15 | 8
Not completed — Explantation of study device(s) | 78 | 47 | 28 | 21
Not completed — Subject Request | 41 | 17 | 13 | 11
Not completed — Lost to Follow-up | 299 | 103 | 51 | 12

BASELINE CHARACTERISTICS:
Population: All enrolled subjects are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Augmentation | Revision-Augmentation | Primary Reconstruction | Revision-Reconstruction | Total
Number analyzed (Participants) | 1116 | 363 | 225 | 84 | 1788
Age, Customized [Number; unit: participants]
  ≤18 | 0 | 0 | 2 | 0 | 2
  18-21 | 47 | 3 | 7 | 0 | 57
  22-25 | 102 | 12 | 5 | 0 | 119
  26-39 | 566 | 128 | 55 | 8 | 757
  40-49 | 335 | 139 | 67 | 26 | 567
  50-59 | 57 | 63 | 62 | 29 | 211
  60-69 | 8 | 18 | 17 | 14 | 57
  70 & over | 1 | 0 | 10 | 7 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1116 | 363 | 225 | 84 | 1788
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1014 | 338 | 204 | 80 | 1636
  Black | 12 | 7 | 5 | 2 | 26
  Hispanic | 37 | 7 | 10 | 1 | 55
  Asian | 29 | 8 | 1 | 0 | 38
  Indian | 1 | 0 | 1 | 0 | 2
  Other | 22 | 2 | 2 | 1 | 27
  Not Provided | 1 | 1 | 2 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 1116 | 363 | 225 | 84 | 1788

OUTCOME MEASURES:

1. Primary Outcome: Local Complications
Description: Assessment of the safety of the Study Implants is based on the incidence of adverse events through 10 years.
Time Frame: 10 Years
Population: All subjects are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Augmentation | Revision-Augmentation | Primary Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 1116 | 363 | 225 | 84
Participants
  Breast Pain | 12 | 7 | 8 | 2
  Baker grade III/IV Capsular Contracture | 120 | 39 | 27 | 9
  Rupture | 42 | 9 | 7 | 5
  Explantation with or without replacement for either cosmetic, medical, or surgical reasons | 151 | 79 | 73 | 36

2. Secondary Outcome: Satisfaction Determined by Patients
Description: Assessment of the effectiveness of Study Implants based on patient satisfaction using a 5-point scale where 1=strongly agree to 5= strongly disagree. The patient satisfaction measures through 10 years provided in the table below are based on questionnaire responses of "Strongly Agree" and "Agree."
Time Frame: 10 Years
Population: All patients that completed the Patient Satisfaction survey at Year 10.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Augmentation | Revision-Augmentation | Primary Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 614 | 176 | 91 | 26
Participants
  Patient thinks her breast implants make her look healthy. | 414 | 110 | 58 | 20
  Patient thinks her breast implants make her look normal. | 444 | 121 | 68 | 22
  Patient thinks her breast implants make her feel more feminine. | 549 | 153 | 70 | 24
  Patient thinks her breast implants make her feel more sensual. | 504 | 141 | 57 | 17
  Patient thinks her breast implants make her clothes feel better. | 482 | 138 | 65 | 23
  Patient thinks her breast implants make her feel more attractive. | 525 | 145 | 64 | 21
  Patient thinks her breast implants make her feel better about herself. | 469 | 137 | 63 | 22
  Patient thinks her breast implants improve her family life. | 118 | 29 | 18 | 10
  Patient thinks her breast implants improve her social life. | 178 | 47 | 26 | 12
  Patient thinks her breast implants improve her daily relations with husband or partner. | 295 | 79 | 32 | 13
  Patient thinks her breast implants improve her sex life. | 319 | 85 | 31 | 9

ADVERSE EVENTS:
Time Frame: Baseline (Surgery) to 10 Years
Arm/Group | Primary Augmentation | Revision-Augmentation | Primary Reconstruction | Revision-Reconstruction
All-Cause Mortality (participants affected / at risk) | 10/1116 | 4/363 | 15/225 | 8/84
Serious Adverse Events (participants affected / at risk) | 0/1116 | 0/363 | 0/225 | 0/84
Other Adverse Events (participants affected / at risk) | 360/1116 | 122/363 | 100/225 | 45/84
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Augmentation (N=1116) | Revision-Augmentation (N=363) | Primary Reconstruction (N=225) | Revision-Reconstruction (N=84)
Asymmetry (Surgical and medical procedures) | 19 | 9 | 22 | 11
Capsular Contracture(Baker Grade II) (Skin and subcutaneous tissue disorders) | 132 | 41 | 27 | 16
Capsular Contracture (Baker Grade III/IV) (Skin and subcutaneous tissue disorders) | 120 | 39 | 27 | 9
Implant Malposition (Surgical and medical procedures) | 26 | 15 | 9 | 7
Infection (Infections and infestations) | 9 | 5 | 11 | 1
Nipple Sensation Changes (Skin and subcutaneous tissue disorders) | 54 | 13 | 4 | 1
Explantation with or without replacement (Surgical and medical procedures) | 151 | 79 | 73 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-08-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT00905645/Prot_SAP_000.pdf